CLINICAL TRIAL: NCT00728585
Title: A Group-Wide Double-Blind Randomized Placebo-Controlled Trial of Palifermin to Prevent Chemotherapy and/or Radiotherapy Induced Oral Mucositis in Children Undergoing Autologous or Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Palifermin in Preventing Oral Mucositis Caused by Chemotherapy and/or Radiation Therapy in Young Patients Undergoing Stem Cell Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ACCL0521; NCI-2009-00329 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000588622; ACCL0521 (Other: Childrens Oncology Group); ACCL0521 (Other: DCP); U10CA095861 (NIH)
Record Dates: First submitted 2008-08-05; First posted 2008-08-06 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2013-04

CONDITIONS: Gastrointestinal Mucositis; Malignant Neoplasm
MeSH Terms: conditions — Mucositis; Neoplasms | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (palifermin) (Experimental): Patients receive palifermin IV once daily for 3 days prior to chemotherapy and/or radiotherapy in the absence of unacceptable toxicity. Patients then receive palifermin IV on days 0, 1, and 2 after autologous or allogeneic hematopoietic stem cell transplantation.
  Interventions: Drug: Palifermin
- Arm II (placebo) (Placebo Comparator): Patients receive placebo IV once daily for 3 days prior to chemotherapy and/or radiotherapy in the absence of unacceptable toxicity. Patients then receive placebo IV on days 0, 1, and 2 after autologous or allogeneic hematopoietic stem cell transplantation.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Palifermin — Given IV
  Other Names: Growth Factor, Recombinant Human Keratinocyte; Kepivance; Keratinocyte Growth Factor, Recombinant Human; Recombinant Human Keratinocyte Growth Factor; rhKGF; rhu Keratinocyte Growth Factor
  Arms: Arm I (palifermin)
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial is studying palifermin to see how well it works compared with a placebo in preventing oral mucositis caused by chemotherapy and/or radiation therapy in young patients undergoing stem cell transplant. Palifermin may help relieve or prevent oral mucositis caused by chemotherapy and radiation therapy in young patients undergoing stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare whether palifermin versus placebo administered to pediatric patients three days prior to conditioning and three days after autologous or allogeneic hematopoietic stem cell transplantation (HSCT) is associated with a reduction in the incidence of WHO grade 3 or 4 oral mucositis.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of palifermin. II. To evaluate the long-term effects of palifermin on disease outcome and survival.

III. To compare the incidence, total dose, and duration of parenteral opioid analgesic use (morphine equivalents), and incidence and duration of total parenteral nutrition (TPN) administration in patients treated with these regimens.

IV. To compare the incidence of febrile neutropenia and invasive bacterial infections in patients treated with these regimens.

TERTIARY OBJECTIVES:

I. To determine whether palifermin versus placebo reduces the incidence of WHO grade 3 or 4 oral mucositis among allogeneic HSCT pediatric patients receiving methotrexate as graft-versus-host disease (GVHD) prophylaxis.

II. To determine whether palifermin versus placebo reduces acute and chronic GVHD after allogeneic HSCT.

III. To describe health care utilization (hospitalization duration, and administration of antibiotics, TPN, nasogastric-, nasojejunal- or gastrostomy-administered enteral nutrition, and blood products) in pediatric patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to age in years (1 to 2 vs 3 to 11 vs 12 to 16), type of hematopoietic stem cell transplantation (HSCT) (autologous vs allogeneic), conditioning regimen (either total-body irradiation [TBI] or melphalan vs neither TBI nor melphalan). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive palifermin IV once daily for 3 days prior to chemotherapy and/or radiotherapy in the absence of unacceptable toxicity. Patients then receive palifermin IV on days 0, 1, and 2 after autologous or allogeneic HSCT.

ARM II: Patients receive placebo IV once daily for 3 days prior to chemotherapy and/or radiotherapy in the absence of unacceptable toxicity. Patients then receive placebo IV on days 0, 1, and 2 after autologous or allogeneic HSCT.

Blood samples are collected at baseline, 32 days, and 100 days after HSCT to evaluate the immunogenicity of palifermin. Oral mucositis is assessed at baseline, daily for 8 days prior to and 32 days after HSCT, or until oral mucositis has resolved by the WHO Mucositis Scale, Oral Mucositis Assessment Scale (OMAS), modified Walsh mucositis scale, Oral Mucositis Daily Questionnaire (OMDQ), and the pain categorical rating scale.

After completion of HSCT, patients are followed periodically for up to 10 years.

ELIGIBILITY:
Criteria:

* Patients undergoing myeloablative autologous or allogeneic hematopoietic stem cell transplantation (HSCT) for any indication
* Any type of myeloablative HSCT conditioning regimen allowed
* Patients undergoing allogeneic HSCT may undergo 1 of the following types of donor stem cells:

  1. HLA-matched sibling or parent
  2. Partially matched family donor (mismatched for a single HLA locus [class I])
  3. Fully matched unrelated marrow or peripheral blood stem cell donor
  4. HLA-matched or partially mismatched (at least 4 of 6 match) cord blood (class I or II)
* Fertile patients must use effective contraception
* No HIV positivity
* No known sensitivity to any E. coli-derived products

  1. Known grade 1 to 2 allergic reactions to asparaginase allowed
  2. No prior grade 3-4 allergies to asparaginase or pegaspargase
* More than 30 days since prior and no concurrent treatment with any of the following therapies:

  1. Oral cryotherapy
  2. Glutamine as an oral supplement
  3. Traumeel
  4. Gelclair
  5. Oral vancomycin paste
  6. Low-level laser therapy
  7. An investigational product or device in another clinical trial
* No prior palifermin or other keratinocyte growth factors
* No other concurrent cytotoxic drugs for conditioning or graft-vs-host disease prophylaxis (intrathecal methotrexate or cytarabine for CNS involvement allowed)
* Not pregnant or nursing

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-03-13 (Actual); Primary Completion 2009-05-08 (Actual)

PRIMARY OUTCOMES:
Incidence of WHO grade 3 or 4 oral mucositis | Up to day 32
  The incidence of WHO grade 3 or 4 mucositis, the palifermin and placebo groups, will be compared using a generalized Cochran-Mantel-Haenszel method for general association as the primary analysis. In addition, this outcome will be examined using a logistic regression model; both approaches will account for the randomization strata. Potential confounders will be examined using multiple logistic regression models.

SECONDARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities of palifermin according to using Common Terminology Criteria for Adverse Events (CTCAE) v 3.0 | Up to 100 days post-HSCT
  Incidence of adverse events and laboratory abnormalities in the palifermin and placebo groups will be summarized for all study participants who receive at least one dose of study medication and also separately for autologous and allogeneic HSCT recipients using descriptive statistics. Time to neutrophil engraftment (first day of ANC 500/mm^3 for at least 2 consecutive days) will be examined in the palifermin and placebo groups and compared using the stratified log rank test. The incidence of serum anti-palifermin antibody formation will be summarized using descriptive statistics.
Long-term effects of palifermin on disease outcome and survival | Up to 10 years
  Long-term outcomes (progression free survival, overall survival and second malignancies) will be examined using Kaplan-Meier and cumulative incidence curves and the compared using the stratified log rank test. These outcomes will be summarized among all study participants and also separately for autologous and allogeneic HSCT recipient.
Duration of WHO grade 3 or 4 oral mucositis | Up to day 32
  Duration of grade 3 or 4 oral mucositis, duration of total parenteral nutrition (TPN) administration and total dose of parenteral opioid analgesic will be compared between groups using a stratified Wilcoxon test. Severity of mucositis according to the Oral Mucositis Assessment Scale (OMAS), modified Walsh mucositis scale, pain categorical rating scale and Oral Mucositis Daily Questionnaire (OMDQ) scales will be compared between groups using the area under the curve (AUC).
Daily OMAS scores | Up to day 32
  The AUC will be compared between groups using a stratified Wilcoxon test, in which stratum-specific rank tests are computed and then summed to obtain a combined test.
Daily modified Walsh mucositis scores | Up to day 32
  The AUC will be compared between groups using a stratified Wilcoxon test, in which stratum-specific rank tests are computed and then summed to obtain a combined test.
Daily pain categorical rating scales | Up to day 32
  The AUC will be compared between groups using a stratified Wilcoxon test, in which stratum-specific rank tests are computed and then summed to obtain a combined test.
Daily OMDQ | Up to day 32
  The AUC will be compared between groups using a stratified Wilcoxon test, in which stratum-specific rank tests are computed and then summed to obtain a combined test.
Incidence, total dose, and duration of parenteral opioid analgesic use (morphine equivalents) | Up to day 32
  Incidence of parenteral opioid analgesic use TPN administration will be compared between groups using a generalized Cochran- Mantel-Haenszel test.
Incidence and duration of total parenteral nutrition administration | Up to day 32
  Incidence of parenteral opioid analgesic use TPN administration will be compared between groups using a generalized Cochran- Mantel-Haenszel test. If subjects are still receiving parenteral opioid analgesia or TPN on day 32, the subsequent stop date also will be collected.
Incidence of febrile neutropenia and invasive bacterial infections | Up to day 32
  The incidence of febrile neutropenia and invasive bacterial infections will be compared using a generalized Cochran-Mantel-Haenszel test.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, Principal Investigator — Children's Oncology Group